CLINICAL TRIAL: NCT00599014
Title: The Atlanta Cardiomyopathy Consortium
Brief Title: Heart Failure Study: The Atlanta Cardiomyopathy Consortium
Acronym: TACC
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Javed Butler, MD, Professor of Medicine, Emory University
Other Study IDs: IRB00005380
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Results first posted 2014-01-01 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-08

CONDITIONS: Heart Failure
Keywords: Cardiomyopathy, heart failure, DNA,; echocardiography, messenger RNA, natural history
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for DNA/RNA/Proteomics analysis and Urine for proteomic analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
Heart failure is a very common cause of hospital admission and there are half a million new cases diagnosed each year in the United States. While some important progress has been made over the last two decades for the treatment of heart failure, there still remains a critical need for further advances in our understanding of this disease in order to significantly improve patient outcomes. Large numbers of heart failure patients need to be studied over time to allow scientists to investigate those factors that influence the responses to therapy.

DETAILED DESCRIPTION:
In this study information will be collected on patients with heart failure and their progress and outcomes will be followed over time. The aim is to understand the natural history, risk factors for improvement or progression, and determinants of response to therapy for heart failure. Of interest are many aspects of heart failure including genetic influences, quality of life issues, how individuals cope with feelings about having heart disease, and how they manage their day-to-day symptoms etc.. A database will be created of approximately 1,000 heart failure patients from Emory, Emory University Hospital Midtown, Wesley Woods, Grady, and the VA Medical Center.

This is strictly an observational study and subjects will not be receiving any experimental therapy nor will their routine medical care be affected in any way. Data to be collected includes:

1. Medical history of the patient
2. Medical history on the patient's family
3. Survey data including health behaviors & psychosocial variables
4. Blood & urine samples
5. EKG
6. Six minute Walk Test
7. Hand grip strength

After collecting data, a variety of statistical tests will be run to analyze factors that influence heart failure patients' responses to treatment. The results of this analysis will be used to optimize therapy for future heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and over
* Sex: Both
* Ethnic Origin: All
* Diagnosis required to participate: Clinical diagnosis of systolic or diastolic heart failure

Exclusion Criteria:

* Congenital heart disease
* Previous heart transplantation
* No primary infiltrative disease i.e. amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiology and general medicine clinics; Inpatients from cardiology services
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2007-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javed Butler, MD, MPH, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Center for Heart Failure at EUH Midtown, 4th Floor, 550 Peachtree Street, Atlanta, Georgia
  - The Emory Clinic, Bldg A., 2nd Floor, 1365 Clifton Road, NE, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were stable patients with heart failure. They were recruited during one of their visits to heart failure clinics. The recruitment period started in November 2007 until December 2010. This was an observational study with no interventions.
Pre-assignment Details: All patients willing to participate to the study were enrolled. Because this was an observational study, no patients with heart failure (ischemic and non-ischemic) were excluded from participation. Only patients with congenital and infiltrated etiologies were not eligible for the study.
Groups:
- Patients With Heart Failure: All stable patients with heart failure willing to participate were enrolled to be followed-up for 5 years
Period: Overall Study
Arm/Group | Patients With Heart Failure
Started | 335
Completed | 335
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Heart Failure
Number analyzed (Participants) | 335
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 300
  >=65 years | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134
  Male | 201
Region of Enrollment [Number; unit: participants]
  United States | 335

OUTCOME MEASURES:

1. Primary Outcome: Death, Heart Transplant, Left Ventricular Assist Device Implantation
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Patients With Heart Failure
Number analyzed (Participants) | 335
participants | 35

2. Secondary Outcome: Hospitalization
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Patients With Heart Failure
Number analyzed (Participants) | 335
participants | 84

ADVERSE EVENTS:
Description: Adverse Events were not collected or observed as part of this observational study.
Arm/Group | Patients With Heart Failure
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Long baseline visit with several questionnaires to be completed made more difficult for the patients to be enrolled. Adverse Events data was not collected as part of this observational registry.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes